CLINICAL TRIAL: NCT05105763
Title: Biofeedback Gait Retraining for Stiff Knee Gait Correction: Multi-joint Adaptation in Children and Young Adults With Brain Injury
Brief Title: Biofeedback Gait Retraining for Stiff Knee Gait Correction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: Children's Specialized Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: R-1084-19
Record Dates: First submitted 2021-09-29; First posted 2021-11-03 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Brain Injury
Keywords: stiff knee gait; biofeedback
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: A counterbalanced repeated measures design will be used in this study to examine the adaptation of children and young adults with brain injury who have SKG to two types of feedback training: feedback training on the knee alone (Condition B) and sequential switched feedback training on the knee and the hip (Condition A). The participants will participate in treadmill training twice with a 2-weeks washout period between the two visits and will receive the two training conditions in different orders. Ten participants will be alternately allocated to two subgroups according to the sequence they are recruited to the study. In the end, the investigators will have five participants in Subgroup 1 and the other five participants in Subgroup 2. Participants in Subgroup 1 will first undergo Condition B in the first visit and then Condition A in the second visit, while participants in Subgroup 2 will start with Condition A in the first visit and then undergo Condition B in the second visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- feedback training on single joint first (Other): Participants in Subgroup 1 will first undergo Condition B in the first visit and then Condition A in the second visit.
  Interventions: Other: Sequential switched feedback training on the knee and the hip (Condition A); Other: Feedback training on the knee alone (Condition B)
- sequential feedback training on multi-joint first (Other): Participants in Subgroup 2 will start with Condition A in the first visit and then undergo Condition B in the second visit.
  Interventions: Other: Sequential switched feedback training on the knee and the hip (Condition A); Other: Feedback training on the knee alone (Condition B)

INTERVENTIONS:
Other: Sequential switched feedback training on the knee and the hip (Condition A) — Condition A will include four 6-mins training blocks: 2-mins knee joint feedback-on, 2-mins hip joint feedback-on, and 2-mins feedback-off. Training with feedback on will occur as follows: The subject will walk on the treadmill and try to achieve the target hip and/or knee flexion pattern shown on the feedback interface. Training with feedback off will occur as follows: The subject will walk on the treadmill and try to maintain the pattern without any form of visual or verbal feedback.
Other: Feedback training on the knee alone (Condition B) — Condition B will include four 6-mins training blocks: 4-mins knee joint feedback-on and 2-mins feedback-off. Training with feedback on will occur as follows: The subject will walk on the treadmill and try to achieve the target hip and/or knee flexion pattern shown on the feedback interface. Training with feedback off will occur as follows: The subject will walk on the treadmill and try to maintain the pattern without any form of visual or verbal feedback.

SUMMARY:
The research team has developed a visual kinematic biofeedback system which is designed to help children with hemiplegic cerebral palsy (CP) correct a pattern of reduced knee extension in terminal swing and early stance. The system provides real-time feedback on the knee angle pattern during walking on a treadmill. From a pilot study on children with CP, the investigators observed that when the system was used in children who have stiff knee gait (SKG), training with knee feedback alone could lead to an increase in hip flexion which in turn led to limited normalization of the knee pattern through the whole gait cycle. This study, funded by the NIDILRR Switzer grant (PI: X Liu, Ph.D.), seeks to address the question of whether a training design with feedback on both the knee and hip joints would reduce this tendency to generate unintended changes in hip joint motion, and in doing so also improve convergence to the intended knee joint pattern. This study will test ten children and young adults with brain injury who have SKG and examine their short term adaptations to two types of kinematic feedback training: feedback training on the knee alone (condition B) and sequential switched feedback training on the knee and the hip (condition A). An additional sensor placed on the pelvis will be added to the current feedback system for measurement and feedback on the hip joint angle. Software enhancements will also be made with methods that will allow study and description of adaptations in measures of inter-limb symmetry during training. The participants will visit twice with a 2-week washout period between the two visits. Five participants will first undergo condition B in the first visit and then condition A in the second visit, while the other five participants will start with condition A in the first visit and then undergo condition B in the second visit. To compare the effects of the conditions on normalizing the joint angle trajectories, the knee and hip kinematics will be collected and analyzed in both the conditions. To investigate the coordination of lower limb segments under feedback training, relative phase measures will be analyzed on the hip and the knee. To examine whether participants adapt to the feedback retraining in terms of improvement in gait quality, symmetry ratios will be analyzed.

DETAILED DESCRIPTION:
Participant characteristics

This study will recruit 10 participants according to the inclusion and exclusion criteria.

System development

In order to measure the quantitative change in hip joint angle online, an additional sensor will be placed on the pelvis segment (overlying the sacrum between the posterior superior iliac spines) and added to the current feedback system. Totally four sensors will be used, including the sensors on the pelvis, thigh, shank, and heel. The hip flexion angle will be calculated from pelvis and thigh sensors. The knee flexion angle will be calculated from thigh and shank sensors, while the heel sensor signal is monitored to isolate strides by detecting contact of the foot with the support surface. To help subjects easily recognize which joint the feedback is cueing for, different backgrounds is selected for the feedback interface for the hip joint and knee joint, respectively. Gait patterns will be video recorded in a sagittal view of the lower extremities. In order to test gait asymmetry by symmetry ratio (dividing the smaller value by the larger value between trained and untrained lower limbs), stance phase duration (% gait cycle) from heel strike to toe off will be identified by motion capturing system with reflective markers. Reflective markers will be placed on the ankles and shoes (fifth metatarsal, heel, rearfoot along the line from heel to toe and below the ankle) on both sides to measure the heel down and toe off events.

Biofeedback gait retraining protocol

Feedback training on the knee alone (Condition B) will include four 6-mins training blocks: 4-mins knee joint feedback-on and 2-mins feedback-off. Sequential switched feedback training on the knee and the hip (Condition A) will include four 6-mins training blocks: 2-mins knee joint feedback-on, 2-mins hip joint feedback-on, and 2-mins feedback-off. Subjects will wear their comfortable footwear and daily used bracing/orthotic devices during the training sessions. Totally four inertial sensors (MTw, Xsens, Netherlands) will be placed separately on the pelvis, anterior thigh, posterior shank and the heel of the paretic lower limb. For calibration purpose, the subject will first stand in his/her natural standing posture and then stand with the knee (weaker side) flexed at 60 degree adding to the knee angle in the natural standing posture. Prior to training, a treadmill walking trial with comfortable speed will be recorded as the baseline trial. After the baseline trial, a 3 minute practice trial will allow interactive demonstration and practice with the goal that the subject has a clear understanding of the task and how to interpret the feedback. In both the two training conditions, subjects will have 3 mins sitting rest between two consecutive blocks to reduce fatigue.

ELIGIBILITY:
Inclusion Criteria:

* age 7 to 21;
* has SKG
* diagnosed with brain injury including but not limited to Cerebral Palsy, Stroke,Traumatic Brain Injury;
* ability to walk on a treadmill without assistive devices based on parent/guardian report and/or treatment history;
* the cognitive development is at the level needed to: understand and follow instructions, answer questions, be able to understand the purpose of the study and the activities involved.

Exclusion Criteria:

* Botulinum toxin treatment less than 16 weeks before initiation of the study
* Recent or concurrent treatment that might interfere with the study.

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-10-30 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-09-29 (Estimated)

PRIMARY OUTCOMES:
Root mean square error of the knee flexion angle | immediate after the first training session
  The root-mean-square error of the knee flexion angle (RMSE_KF) will be calculated between the measured and target knee flexion angles in the last ten strides of the last trial with feedback off in each training session.
Root mean square error of the knee flexion angle | immediate after the second training session
  The root-mean-square error of the knee flexion angle (RMSE_KF) will be calculated between the measured and target knee flexion angles in the last ten strides of the last trial with feedback off in each training session.
Peak knee flexion angle | immediate after the first training session
  The Peak knee flexion angle (PKF) is the mean maximum knee flexion angles in the last ten strides of the last trial with feedback off.
Peak knee flexion angle | immediate after the second training session
  The Peak knee flexion angle (PKF) is the mean maximum knee flexion angles in the last ten strides of the last trial with feedback off.
Peak hip flexion angle | immediate after the first training session
  The Peak hip flexion angle (PHF) is the mean maximum knee flexion angles in the last ten strides of the last trial with feedback off.
Peak hip flexion angle | immediate after the second training session
  The Peak hip flexion angle (PHF) is the mean maximum knee flexion angles in the last ten strides of the last trial with feedback off.
Minimum relative phase angle between hip and knee | immediate after the first training session
  Minimum relative phase angle between hip and knee is the minimum difference in phase angle between hip and knee. Phase angle is computed as the inverse tangent of angular velocity divided by angular displacement.
Minimum relative phase angle between hip and knee | immediate after the second training session
  Minimum relative phase angle between hip and knee is the minimum difference in phase angle between hip and knee. Phase angle is computed as the inverse tangent of angular velocity divided by angular displacement.
Symmetry ratio of the stance phase | immediate after the first training session
  The symmetry ratio is calculated by dividing the smaller value by the larger value (trained vs. untrained lower limbs) of the stance phase time (% gait cycle). This results in a value between 0.0 and 1.0, with values closer to 1.0 indicating greater symmetry.
Symmetry ratio of the stance phase | immediate after the second training session
  The symmetry ratio is calculated by dividing the smaller value by the larger value (trained vs. untrained lower limbs) of the stance phase time (% gait cycle). This results in a value between 0.0 and 1.0, with values closer to 1.0 indicating greater symmetry.

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Liu, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No